CLINICAL TRIAL: NCT02174536
Title: A Double Blind Randomized Study Using Placenta Derived Decidual Stromal Cells for Hemorrhagic Cystitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Olle Ringdén, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSCHC002
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Hemorrhagic Cystitis; Stem Cell Transplantation; Decidual Stromal Cells
MeSH Terms: conditions — Cystitis, Hemorrhagic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Decidual Stromal cell therapy (Active Comparator): Decidual stromal cell therapy (approximately 1x10^6 cells/kg) for hemorrhagic cystitis in addition to Misoprostol therapy (0,2mg, 3 times/day) on two occasions at weekly intervals.
  Interventions: Biological: Decidual stromal cells
- Placebo (Placebo Comparator): Receives placebo (masked i.v. infusion, same amount as an infusion of decidual stromal cells) in addition to Misoprostol therapy (0,2mg, 3 times/day).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Decidual stromal cells — Decidual stromal cells (approximately 1x10^6 cells/kg) will be infused intravenously.
  Arms: Decidual Stromal cell therapy
Biological: Placebo
  Arms: Placebo

SUMMARY:
A prospective double blind randomized study comparing placenta derived decidual stromal cells with placebo for hemorrhagic cystitis after allogeneic hematopoietic cell transplantation. It is hypothesized that the decidual stromal cell therapy will be superior to placebo.

DETAILED DESCRIPTION:
Patients with grade 2-4 hemorrhagic cystitis will be randomized to receive either decidual stromal cell therapy at approximately 1x106 cells/kg or placebo on two occasions at weekly intervals. Patients not responsive within 2 weeks will receive decidual stromal cells at approximately 1x106 cells/kg openly.

ELIGIBILITY:
Inclusion Criteria:

* Hemorrhagic cystitis grade 2-4
* Receives Misoprostol therapy

Exclusion Criteria:

* Patients with urinary urge without macroscopic hematuria or clots

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Days to disappearence of macroscopic hematuria or clots | 1 month after inclusion
  Each day, patients fill out a form were they state whether they have macroscopic hematuria or not.

SECONDARY OUTCOMES:
Time to disappearance of pain or urges | 1 month after inclusion
Time to disappearance of microscopic hematuria | 1 month after inclusion
  Each day patients, with the help of a urinary test stick, fill out a form were they state whether they have microscopic hematuria or not.
Transplant related mortality | 1 year after inclusion
  All mortality except relapse
Incidence of severe infections | 1 year after inclusion
  Incidence of severe bacterial, viral or fungal infections.
Incidence of graft versus host disease | One year after inclusion
Overall actuarial survival | Actuarial

CONTACTS AND LOCATIONS:
Overall Officials: Olle Ringdén, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden